CLINICAL TRIAL: NCT01722396
Title: The Pharmacogenetics of Vitamin D Supplementation in Tuberculosis
Brief Title: Pharmacogenetics of Vitamin D Supplementation in Tuberculosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Heart of England NHS Trust (Other)
Responsible Party: Principal Investigator, Alice Turner, Clinician Scientist and Honorary Consultant Physician, University of Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG-10-179
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D (Experimental)
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D

SUMMARY:
Previous studies of vitamin D supplementation have suggested there may be differences in response between individuals. This study is an open label study of vitamin D supplementation in patients with active or latent tuberculosis in which active disease patients take 100000units of vitamin D every 8 weeks during their tuberculosis treatment. Genotyping for relevant vitamin D pathway polymorphisms will be carried out and related to clinical and ex vivo markers of vitamin D response. Latent patients will only be studied for vitamin D response ex vivo. Our hypothesis is that response to vitamin D in both monocytes and T cells will be related to polymorphisms in the DBP gene, and that this may relate to clinical response in terms of post supplementation vitamin D level.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or above
* Microbiologically or histologically confirmed active tuberculosis
* Clinically confirmed latent tuberculosis

Exclusion Criteria:

1. Patients being managed with regimes outside standard NICE guidance
2. Drug resistant MTb
3. HIV positive
4. Known intolerance of vitamin D
5. Sarcoidosis
6. Hyperparathyroidism or nephrolithiasis
7. Taking vitamin D supplementation in the two months preceding enrolment
8. Baseline serum corrected calcium >2.65 mmol/L
9. Current haemodialysis
10. Children, pregnant or breastfeeding individuals
11. Concomitant benzothiadiazine derivative, cardiac glycoside, carbamazepine, phenobarbital, phenytoin, primidone or long-term immunosuppressant therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in post supplementation vitamin D level | 8,16 and 24 weeks

SECONDARY OUTCOMES:
Ex vivo responses of monocytes to vitamin D | 0 and 8 weeks
Ex vivo responses of T cells to vitamin D | 0 and 8 weeks

OTHER OUTCOMES:
Serum levels of inflammatory markers | 0, 8 , 16 and 24 weeks
Serum levels of calcium | 0,8, 16 and 24 weeks
TB score | 0,8.16 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alice Turner, Principal Investigator — University of Birmingham
Locations (1):
- Heart of England NHS Trust, Birmingham, West Midlands, United Kingdom